CLINICAL TRIAL: NCT04511559
Title: Methylation Analysis of Circulating Tumor DNA in Early Diagnosis and Prognostic Stratification in Patients With Gastric Cancer
Brief Title: Methylation Analysis of Circulating Tumor DNA in Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-DL-202001
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Stomach Neoplasms; Circulating Tumor DNA
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- chronic gastritis: This group will include 80 patients with chronic gastritis and the diagnoses will be based on the British Society of Gastroenterology guidelines.
  Interventions: Diagnostic Test: Circulating Tumor DNA Methylation Sequencing; Diagnostic Test: tissue DNA Methylation Sequencing
- Moderate to severe atrophy/intestinal metaplasia/: This group will include 80 patients with Moderate to severe atrophy/intestinal metaplasia/ and the diagnoses will be based on British Society of Gastroenterology guidelines.
  Interventions: Diagnostic Test: Circulating Tumor DNA Methylation Sequencing; Diagnostic Test: tissue DNA Methylation Sequencing
- gastric cancer: This group will include 380 patients with gastric cancer and the diagnoses will be based on British Society of Gastroenterology guidelines.
  Interventions: Diagnostic Test: Circulating Tumor DNA Methylation Sequencing; Diagnostic Test: tissue DNA Methylation Sequencing

INTERVENTIONS:
Diagnostic Test: Circulating Tumor DNA Methylation Sequencing — Whole blood collection through venipuncture. DNA methylation levels by deep sequencing.
Diagnostic Test: tissue DNA Methylation Sequencing — Isolate DNA from tissue samples from subjects. DNA methylation levels by deep sequencing.

SUMMARY:
The primary purpose of this trial is to describe the profile of ctDNA methylation in gastric cancer. The second purpose is to demonstrate the correlation between the plasma ctDNA methylation status and the diagnosis and prognosis of patients with early and intermediate stage gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer represents one of the common malignant tumors in China, with high incidence and mortality rates. Surgery is the conventional treatment option for early and intermediate stage gastric cancer, but the diagnosis in the early stage of gastric cancer remains a challenge to clinical practitioners. Circulating tumor DNA (ctDNA) is tumor-derived fragmented DNA with an average size of 166 bp, mixed with cell-free DNA (cfDNA) of other sources in blood circulation. ctDNA is reflecting the most up-to-date status of the tumor genome. Hence, it is considered as a novel biomarker for tumors, which can be qualitative, quantitative, and used for disease monitoring. This study is designed to evaluate the potential clinical utility of circulating tumor DNA (ctDNA) as a clinical index in the diagnosis and prognosis of gastric cancer. The primary purpose of this trial is to describe the profile of ctDNA methylation in gastric cancer. The second purpose is to demonstrate the correlation between the plasma ctDNA methylation status and the diagnosis and prognosis of patients with early and intermediate stage gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is scheduled to undergo an endoscopy because of medical indications.
2. The subject must have personally signed and dated the patient informed consent form indicating that he/she has been informed of all pertinent aspects of the study.
3. The subject must be willing and able to comply with all study procedures.

Exclusion Criteria:

1. The subject who is unable to undergo gastroscopy.
2. The subject with previous total or partial gastrectomy.
3. The subject has other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may interfere with the interpretation of study results and in the judgment of the investigator would make the subject unsuitable for entry into the study.
4. The subject is unwilling or unable to provide signed informed consent.
5. The subject who is pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred to the participating study sites for upper GI endoscopy for standard clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Analysis ctDNA methylation status and its Correlation to early diagnosis and prognostic evaluation of gastric cancer. | 1-2 years
  We will develop the linear model and a threshold value differentiating gastric cancer from control based on the 100 patient training set.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Diaz LA Jr, Bardelli A. Liquid biopsies: genotyping circulating tumor DNA. J Clin Oncol. 2014 Feb 20;32(6):579-86. doi: 10.1200/JCO.2012.45.2011. Epub 2014 Jan 21. PMID 24449238
- [Background] Kilgour E, Rothwell DG, Brady G, Dive C. Liquid Biopsy-Based Biomarkers of Treatment Response and Resistance. Cancer Cell. 2020 Apr 13;37(4):485-495. doi: 10.1016/j.ccell.2020.03.012. PMID 32289272
- [Background] Gao Y, Zhang K, Xi H, Cai A, Wu X, Cui J, Li J, Qiao Z, Wei B, Chen L. Diagnostic and prognostic value of circulating tumor DNA in gastric cancer: a meta-analysis. Oncotarget. 2017 Jan 24;8(4):6330-6340. doi: 10.18632/oncotarget.14064. PMID 28009985